CLINICAL TRIAL: NCT03278301
Title: A Multicenter Post-Market Registry for the Evaluation of the CorPath® GRX System Effectiveness in Percutaneous Coronary Interventions
Brief Title: PRECISION GRX Registry
Status: Completed | Type: Observational
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-001
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Robotic-assisted PCI — The CorPath GRX is intended for use in the remote delivery and manipulation of guidewires and rapid exchange balloon/stent catheters, and remote manipulation of guide catheters during percutaneous coronary intervention (PCI) procedures.

SUMMARY:
To collect data on the routine patterns of use, safety and effectiveness, including the clinical and technical performance of the CorPath GRX System, in the delivery and manipulation of coronary guidewires and stent/balloon catheters, and manipulation of guide catheters during PCI procedures.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multi-center patient registry of the CorPath GRX System to examine its performance during PCI procedures and patient outcomes through 72 hours post-procedure or hospital discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Candidates will be included in the study only if all of the following conditions are met:

1. Age ≥18 years;
2. Patients with coronary artery disease with clinical indication for PCI;
3. Patient deemed appropriate for robotic-assisted PCI; and
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Candidates will be excluded from the study if any of the following conditions are present:

  1. Failure/inability/unwillingness to provide informed consent; or
  2. The investigator determines that the patient or the coronary anatomy is not suitable for robotic-assisted PCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease and with a clinical indication for PCI.
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2017-08-27 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Discharge or 72 hours post intervention, whichever comes first.
  Less than 30% residual stenosis (visual estimate) post PCI in the lesion(s) treated with the CorPath GRX System, without in-hospital major adverse coronary events (MACE).
Technical Success | Procedure
  Defined as successful completion of the robotic-assisted PCI absent unplanned conversion to manual for guidewire or balloon/stent catheter inability to navigate vessel anatomy or poor guide catheter support.

SECONDARY OUTCOMES:
Overall Procedure Time | Procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
PCI Procedure Time | Procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Fluoroscopy Time | Procedure
  Total Fluoroscopy Time during procedure will be captured.
Patient Radiation Exposure | Procedure
  DAP (dose-area-product) and cumulative dose/air kerma as recorded during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ehtisham Mahmud, MD, Principal Investigator — University of California, San Diego
Locations (20):
- United States (17):
  - UC San Diego Health Sulpizio Cardiovascular Center, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Spectrum Health Hospitals Fred and Lena Meijer Heart Center, Grand Rapids, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - New York-Presbyterian Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - WakeMed Raleigh Campus, Raleigh, North Carolina
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Wellspan York Hospital, York, Pennsylvania
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Health System University Hospital, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Albert Einstein Israelite Hospital, São Paulo, São Paulo, Brazil
- Apex Heart Institute, Ahmedabad, Gujarat, India
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No